CLINICAL TRIAL: NCT00231881
Title: Functional and Molecular Characterisation of Oesophageal Distal Epithelium: Correlations With Acid and Non Acid Reflux
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Other Study IDs: BRD 05-3-H
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2007-04-30 (Estimated); Status verified 2007-04

CONDITIONS: Gastroesophageal Reflux
Keywords: GORD - Oesophageal sensitivity- Oesophageal permeability
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This study aims to characterize the permeability as well as some protein involved in the cell junction in the oesophageal epithelium in patients with GORD symptoms. In addition these patients will be characterized for their reflux especially by pH-impedancemetry, Bilitec and oesophageal acid perfusion test. Correlations between the characteristics of the reflux and the biological results will be calculated.

DETAILED DESCRIPTION:
This study aims to characterize the permeability as well as some protein involved in the cell junction in the oesophageal epithelium in patients with GORD symptoms. In addition these patients will be characterized for their reflux especially by pH-impedancemetry, Bilitec and oesophageal acid perfusion test. Correlations between the characteristics of the reflux and the biological results will be calculated.

ELIGIBILITY:
Inclusion Criteria:

Main inclusion criteria :

* Digestive symptoms suggestive of GORD (heartburn, regurgitation, epigastric pain), or dyspeptic syndrome (nausea, belch, bloating, epigastric discomfort).
* Need of upper GI endoscopy and pH monitoring.
* Normal propagation of oesophageal persitaltic waves (manometry < 6 months).
* Age 18 -70 yrs
* Signed informed consent
* Normal coagulation

Exclusion Criteria:

* Barrett's oesophagus
* Previous oesophageal bleeding
* Need of NSAID treatment.
* Previous sus mesocolic surgery
* Alcool consumption > 40g/d, smoking > 10 cig/j
* Pregnancy or lack of contraceptive disposal, breast feeding.
* Allergy to Xylocaïne

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas Bruley des Varannes, Md, Principal Investigator — Centre Hospitalier et Universitaire de Nantes
Locations (1):
- Nantes University Hospital, Nantes, France